CLINICAL TRIAL: NCT05420233
Title: The CROCO Study: CROhn's Disease COhort Study
Acronym: CROCO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GLSMED Learning Health S.A. (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: The CROCO Study
Record Dates: First submitted 2022-05-25; First posted 2022-06-15 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: Crohn Disease
Keywords: Crohn DII
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients diagnosed with Crohn´s disease within the past 12 months (Other): All patients will undergo MRE in year 1, and this test may not be recommended in all patients. Year 1 MRE is the only procedure that may be performed outside of clinical practice.
  Interventions: Diagnostic Test: MRE

INTERVENTIONS:
Diagnostic Test: MRE — Magnetic Resonance Enterography at year 1 (in some patients)
  Other Names: Magnetic Resonance Enterography

SUMMARY:
The investigators propose to create a prospective Crohn Disease cohort, where patients receiving the most up-to-date therapies with a treat-to-target strategy, will be closely followed to characterize the progression of Crohn Disease by measuring the Lémann Index over time. The goal of the CROCO Study - "Crohn's Disease Cohort Study" is to promote a greater understanding of the long-term evolution of Crohn Disease , to describe prospectively the impact of different therapeutic strategies and develop accurate predictors of bowel disease damage and disability.

DETAILED DESCRIPTION:
Therefore, the investigators designed a prospective, multicentre, study of the clinical course, anatomical progression and treatment of newly diagnosed CD and plan to include 600 patients over a 2-year period. Patients will be followed over 5 years after diagnosis (the date of diagnosis will be the date of the index histopathology describing CD; in special situations where pathology is not available the date of diagnosis will be the date that CD was declared by the physician). A morphological evaluation (LI), using abdominal magnetic resonance, will be performed at 1, 3 and 5 years after diagnosis. Ileocolonoscopy, upper endoscopy and/or pelvic MRI will be included according to disease location. Patients will be treated with standard of care therapy and will be followed for 5 years after diagnosis, with semestrial visits after the Year 1 (LI 1). At each visit, clinical and laboratory markers will be collected. Perianal and abdominal surgeries during follow-up will be registered. The disability index questionnaire will also be recorded every year.

A preliminary requisite is therefore to implement and standardize examination reports and damage definitions used to calculate the LI. To this end, training session, supervised by members of the steering committee, will be held for participating gastroenterologist and radiologists. Based on commented ileocolonoscopy, upper endoscopy abdominal MRI and pelvic MRI, these sessions will highlight how lesions should be characterized and graded accordingly to implement the Lémann Index.

ELIGIBILITY:
INCLUSION CRITERIA

To be eligible all of the following criteria must be met:

* Diagnosis of CD (according to ECCO guidelines) established within the past 12 months;
* Patients able to understand the information provided to them and to give written informed consent for the study;
* Male or female, age > 18 years.

EXCLUSION CRITERIA:

* Patients unwilling or unable to provide informed, written consent;
* Severe underlying medical disorder with an anticipated life expectancy < 2 years;
* Refusal or medical conditions (e.g. Glomerular filtration rate < 30 mL/min) preventing cross-sectional imaging during follow-up;
* Uncertain CD diagnosis;
* Pregnancy (if it is impossible to implement the MRE at one year) or any other reason that makes resonance not feasible throughout the study (eg claustrophobia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Lémann Index Y1 | 1 year after diagnosis
  The Lémann Index (LI) was developed to provide a tool to measure bowel damage in Crohn Disease (CD).
  Descriptive statistics will present quantitative variables as mean and standard deviation or median and interquartile range (depending on their distribution) and qualitative variables as count and percentage.
  Time to event endpoints (such as surgery and hospitalization) will be presented using cumulative incidence in a competing risk framework (with death without surgery as a competing event for time to surgery, for example). Cumulative incidence with its 95%CI will be estimated at meaningful timepoints and association between baseline predictors and time to event endpoint will be assessed using competing risks regression models. Correlation of LI and IBD-DI will be estimated, taking into account the repeated measurements.
  Lémann Index is a continuous variable.
Lémann Index Y3 | 3 years after diagnosis
  The Lémann Index (LI) was developed to provide a tool to measure bowel damage in Crohn Disease (CD).
  Descriptive statistics will present quantitative variables as mean and standard deviation or median and interquartile range (depending on their distribution) and qualitative variables as count and percentage.
  Time to event endpoints (such as surgery and hospitalization) will be presented using cumulative incidence in a competing risk framework (with death without surgery as a competing event for time to surgery, for example). Cumulative incidence with its 95%CI will be estimated at meaningful timepoints and association between baseline predictors and time to event endpoint will be assessed using competing risks regression models. Correlation of LI and IBD-DI will be estimated, taking into account the repeated measurements.
  Lémann Index is a continuous variable.
Lémann Index Y5 | 5 years after diagnosis
  The Lémann Index (LI) was developed to provide a tool to measure bowel damage in Crohn Disease (CD).
  Descriptive statistics will present quantitative variables as mean and standard deviation or median and interquartile range (depending on their distribution) and qualitative variables as count and percentage.
  Time to event endpoints (such as surgery and hospitalization) will be presented using cumulative incidence in a competing risk framework (with death without surgery as a competing event for time to surgery, for example). Cumulative incidence with its 95%CI will be estimated at meaningful timepoints and association between baseline predictors and time to event endpoint will be assessed using competing risks regression models. Correlation of LI and IBD-DI will be estimated, taking into account the repeated measurements.
  Lémann Index is a continuous variable.

CONTACTS AND LOCATIONS:
Overall Officials: Joana T Torres, Phd, Principal Investigator — Luz Saude
Locations (20):
- University Hospital CHU of Liège, Liège, Liège, Belgium
- American Gastroenterology Center, Stróvolos, Cyprus
- IBD Clinical and Research Clinic, ISCARE, Prague, Czechia
- Denmark (2):
  - Hvidovre Hospital, Hvidovre
  - Slagelse Hospital, Slagelse
- France (3):
  - CHU Amiens-Picardie Hôpital Sud, Amiens
  - CHU Estaing Clermont - Ferrand, Clermont-Ferrand
  - Claude Huriez Hospital, Lille University, Lille
- Italy (2):
  - Azienda Ospedaliera di Padova, Padua
  - Ospedale San Raffaele, San Raffaele
- Mater dei hospital, Msida, Malta
- Portugal (3):
  - Hospital Garcia da Orta, Almada, Almada
  - Instituto Portugues de Oncologia de Lisboa, Lisbon, Lisbon District
  - Hospital Beatriz Angelo, Loures, Loures
- Algomed Policlinic, Timișoara, Romania
- Spain (3):
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Galdakao-Usansolo, Galdakao
  - Hospital Alvaro Cunqueiro - Área Sanitária de Vigo, Vigo
- United Kingdom (2):
  - Hull University Teaching Hospitals NHS Trust, Hull
  - St Mark's Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reves J, Buisson A, Burisch J, Arebi N, Ungaro R, Vieujean S, Cravo M, Ellul P, Duricova D, Sebastian S, Rodriguez-Lago I, Ordas I, Kaimakliotis I, Hernandez V, Mocanu I, Nachury M, Goldis A, Fumery M, Conceicao D, Pedersen NK, Guedes AF, Ribeiro R, Bigot N, Mary JY, Lambert J, Colombel JF, Torres J; CROCO Study Group. The CROCO (CROhn's Disease COhort Study) - study design and protocol. Therap Adv Gastroenterol. 2025 Aug 29;18:17562848251362594. doi: 10.1177/17562848251362594. eCollection 2025. PMID 40895198